CLINICAL TRIAL: NCT01603693
Title: Bone Quality and Quantity Following Guided Bone Regeneration With Bio-Oss Alone or Combined With BondBone, Prior to Dental Implant Placement
Brief Title: Bone Quality and Quantity Following Guided Bone Regeneration Prior to Dental Implant Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BioOss-BondBone-HMO-CTIL
Record Dates: First submitted 2012-05-07; First posted 2012-05-22 (Estimated); Last update posted 2017-11-28 (Actual); Status verified 2012-03

CONDITIONS: Resorbed Alveolar Ridge Prior to Dental Implant Insertion
Keywords: Guided bone regeneration; Bio Oss; BondBone; computerized tomography; histological examination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bio-Oss (Experimental): In this arm,GBR will be performed with DBBM (Bio-Oss, Geistlich) in 25 patients.
  Interventions: Device: Bio-Oss (by Geistlich)
- Bio-Oss and BondBone (Experimental): In this arm, GBR will be performed using a combination of DBBM (Bio-Oss, Geistlich) and bi-phasic calcium sulphate (BondBone, Augma) in 25 patients.
  Interventions: Device: Bio-Oss (by Geistlich); Device: BondBone (by Augma)

INTERVENTIONS:
Device: Bio-Oss (by Geistlich) — Guided Bone Regeneration (GBR) will be done with no changes from the common (Dahlin 1988). Patients will be given local anasthesia, full thickness mucoperiosteal flap will be raised to expose the bone area that needs augmentation, bone substitute will be placed over the bony crater and covered with a collagen membrane (Bio-Gide, geistlich, FDA and CE approved). Mucoperiosteal flap will be sutured and patients will be instructed to a check-up routine as accepted after this kind of procedure.
  Other Names: Deproteinized Bovine Bone Mineral
Device: BondBone (by Augma) — Guided Bone Regeneration (GBR) will be done with no changes from the common (Dahlin 1988). Patients will be given local anasthesia, full thickness mucoperiosteal flap will be raised to expose the bone area that needs augmentation, bone substitute will be placed over the bony crater and covered with a collagen membrane (Bio-Gide, geistlich, FDA and CE approved). Mucoperiosteal flap will be sutured and patients will be instructed to a check-up routine as accepted after this kind of procedure.
  Other Names: bi-phasic Calcium-Sulphate
  Arms: Bio-Oss and BondBone

SUMMARY:
Amongst the consequences of missing teeth are change of appearance and difficulties in mastication and speech. Dental implants in the maxilla or mandible provide a common treatment modality by offering anchorage to fixed or removable fixtures. In many cases, the lack of teeth is accompanied by lack of appropriate bone volume in the desired area for dental implant placement. Possible causes for this lack of sufficient bone volume are varied and include earlier bone atrophy, traumatic tooth extraction and bone resorption due to periodontal disease. In such cases, dental implant placement is preceded by alveolar bone augmentation . Guided Bone Regeneration (GBR) is a common bone augmentation technique in which a bulk of bone substitute is placed in the area which needs more volume before placing a dental implant. The bone substitute is covered with an inert membrane and may provide a scaffold and encourage cells from the patient to reach the area and build new bone volume. A common bone substitute in use for that matter is Deproteinized bovine bone mineral (DBBM) which resembles human bone and helps encourage new bone formation. On the contrary its structural stability during placement and early healing is low. Bi-Phasic Calcium-Sulphate is another common bone substitute with easy handling properties and good structural stability during early healing. Its replacement by natural bone contributes to the augmentation process. Although DBBM efficacy in GBR process has been investigated, using DBBM in combination with bi-phasic calcium-sulphate as a binding material during GBR was not examined. This prospective study will examine augmented bone quality and quantity following a GBR procedure with common approved bone substitutes: DBBM (Bio-Oss, Geistlich) alone or in a combination with bi-phasic Calcium-sulphate (BondBone, Augma). The GBR procedures will precede dental implant placement as custom. The quality and quantity of the new formed bone will be assessed by a C.T (computerized tomography) which is done routinely before dental implant placement and by further analyses of bone residues which will follow drilling the dental implant placement site while preparing it (as common).

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women over 18 years of age, eligible for signing
* Edentulus Patients who require a GBR procedure previous to an insertion of a dental implant
* Patients who understand the meaning of the treatment (routine Guided Bone Regeneration and dental implant insertion) and the follow up study, and approves participation in booth of them

Exclusion Criteria:

* Pregnant or nursing women.
* C567890-hildren or non judgemental patients
* Patients with uncontrolled diabetas mellitus, rheumatoid arthritis or osteoporosis.
* Patients with a pathology present near the site of dental implantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2013-02-21 (Actual); Study Completion 2013-02-21 (Actual)

PRIMARY OUTCOMES:
Volume of the new bone formed after a GBR procedure | Volume of the new bone formed after the GBR procedure will be determined up to 7 months after the GBR procedure and before the insertion of dental implants.
  Bone volume obtained following a GBR procedure will be detemined through a comparison of a 3 dimensional analysis of computed tomography images done before and after the GBR procedure.

SECONDARY OUTCOMES:
Bone quality | Bone quality will be assesed through histological analysis that will be carried out at the time of implants insertion (up to 8 months following the GBR procedure).
  The collected bone sample will be subjected to histo-morphometric analysis in order to determine the size, shape and orientation of the bony trabeculae,the size and porosity of the bony cortex in addition to the new bone/ bone substitute ratio.

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Background] Lang NP, Hammerle CH, Bragger U, Lehmann B, Nyman SR. Guided tissue regeneration in jawbone defects prior to implant placement. Clin Oral Implants Res. 1994 Jun;5(2):92-7. doi: 10.1034/j.1600-0501.1994.050205.x. PMID 7918914